CLINICAL TRIAL: NCT05897450
Title: The Effects of TAP Block on Thiol/Disulfide Homeostasis and Pain in Laparoscopic Gynecological Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara Etlik City Hospital (Other Government)
Responsible Party: Principal Investigator, Yusuf Özgüner, Principal Investigator, Ankara Etlik City Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: AnkaraEtlikYusufOzguner002
Record Dates: First submitted 2023-06-01; First posted 2023-06-09 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-06

CONDITIONS: Pain, Postoperative; Oxidative Stress
Keywords: thiol/disulphide homeostasis; TAP block; Laparoscopic Gynecological Surgery
MeSH Terms: conditions — Pain, Postoperative | interventions — Dental Occlusion

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients with TAP block (Active Comparator): After induction of anesthesia, TAP block was applied to the patients under ultrasound guidance.
  Interventions: Other: Transversus abdominis plane (TAP) block
- Patients without TAP block (Other): Local anesthetic infiltration was applied to the trocar sites with the same volume.
  Interventions: Other: Local anesthetic infiltration

INTERVENTIONS:
Other: Transversus abdominis plane (TAP) block — Transversus abdominis plane (TAP) block: injection of a local anesthetic into a region between the internal oblique and transversus abdominis muscles.
  Arms: Patients with TAP block
Other: Local anesthetic infiltration — Local anesthetic infiltration was applied to the trocar sites with the same volume.
  Arms: Patients without TAP block

SUMMARY:
In the study, it was aimed to compare patients who underwent laparoscopic gynecological surgery with and without TAP block in terms of postoperative pain levels and Thiol/Disulfide homeostasis.

DETAILED DESCRIPTION:
Thiols are organic sulphur derivatives containing Sulfhydryl Residues (-SH) in their active regions. Thiols easily react with oxygen containing free radicals to form disulfides. This is a defence mechanism against oxidative stress.7 An automated analysis quantitatively measuring serum native and total thiol, and disulfides has been recently described as a method to determine dynamic Thiol/Disulfide Homeostasis (TDH).The role of dynamic thioldisulfide homeostasis has been increasingly shown in many diseases. There is a growing number of evidences that an abnormal thiol-disulfide homeostasis may play role in the pathogenesis of a variety of diseases such as cardiovascular disease, malignancies, rheumatoid arthritis, chronic kidney disease, and acquired immunodeficiency syndrome.

Laparoscopic gynecological surgery has several advantages when compared to open surgery, including faster postoperative recovery and lower pain scores. However, the possibility of significant postoperative pain remains. Trocar placement, tissue dissection, and pneumoperitoneum formation contribute to postoperative pain in laparoscopic surgery. If this pain is not treated adequately, it can cause an increase in pain levels, nausea and vomiting, and as a result, a decrease in patient comfort and a prolongation of hospitalization. Ultrasound-guided transversus abdominis plane (TAP) block is easy to perform and has recently become a popular technique for reducing postoperative pain after abdominal surgery. It has been reported that it provides effective postoperative analgesia with a decrease in opioid consumption in various open abdominal surgical procedures and contributes to faster patient recovery.

In the study, it was aimed to compare patients who underwent laparoscopic gynecological surgery with and without TAP block in terms of postoperative pain levels and Thiol/Disulfide homeostasis.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have undergone laparoscopic gynecological surgery
* Patients who agreed to participate in the study

Exclusion Criteria:

* Patients who did not agree to participate in the study
* Patients with missing data

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-07-15 (Actual); Primary Completion 2023-12-15 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
Thiol/Disulphide Homeostasis | 5 minutes before induction of anesthesia
  In order to determine thiol / disulphide homeostasis, 5 ml blood samples were taken 2 times from each patient (T1: 5 minutes before induction of anesthesia, T2: at the time of the surgery over).
Thiol/Disulphide Homeostasis | postoperative 24th hour
  In order to determine thiol / disulphide homeostasis, 5 ml blood samples were taken 2 times from each patient (T1: 5 minutes before induction of anesthesia, T2: at the time of the surgery over).

SECONDARY OUTCOMES:
Pain on the Numeric Rating Scale (NRS) | 0 hours postoperatively, 2 hours postoperatively,4 hours postoperatively,8 hours postoperatively,12 hours postoperatively,24 hours postoperatively
  Participants recorded pain rated on the numeric rating scale (NRS) at 6 time points: 0 hours postoperatively, 2 hours postoperatively, 4 hours postoperatively, 8 hours postoperatively, 12 hours postoperatively, 24 hours postoperatively. NRS range was from 0-10 with 0 being no pain and 10 the worst pain possible.

CONTACTS AND LOCATIONS:
Overall Officials: Yusuf Ozguner, Principal Investigator — Ankara Etlik City Hospital
Locations (1):
- Ankara Etlik City Hospital, Ankara, Varlık Mahallesi, Halil Sezai Erkut Caddesi Yenimahalle, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Erel O, Neselioglu S. A novel and automated assay for thiol/disulphide homeostasis. Clin Biochem. 2014 Dec;47(18):326-32. doi: 10.1016/j.clinbiochem.2014.09.026. Epub 2014 Oct 7. PMID 25304913
- [Background] Oksuz M, Abitagaoglu S, Kaciroglu A, Koksal C, Ozturk BY, Erel O, Senat A, Erdogan Ari D. Effects of general anaesthesia and ultrasonography-guided interscalene block on pain and oxidative stress in shoulder arthroscopy: A randomised trial. Int J Clin Pract. 2021 Dec;75(12):e14948. doi: 10.1111/ijcp.14948. Epub 2021 Oct 12. PMID 34614288
- [Background] Baeriswyl M, Kirkham KR, Kern C, Albrecht E. The Analgesic Efficacy of Ultrasound-Guided Transversus Abdominis Plane Block in Adult Patients: A Meta-Analysis. Anesth Analg. 2015 Dec;121(6):1640-54. doi: 10.1213/ANE.0000000000000967. PMID 26397443